CLINICAL TRIAL: NCT01957254
Title: Investigate the Activity of Endotoxin in Patients With Severe Sepsis and Septic Shock
Brief Title: Investigate the Activity of Endotoxin in Severe Sepsis
Status: Terminated | Type: Observational
Why Stopped: The quality of Limulus Amebocyte Lysate (LAL) test was poor.
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201211040RIB
Record Dates: First submitted 2013-07-04; First posted 2013-10-08 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe Sepsis: Patient with severe sepsis

SUMMARY:
Endotoxin is the major mediator of gram-negative bacteria which cause the systemic inflammation and result in microcirculatory dysfunction, and it leads to multiple organ dysfunction and death in patients with severe sepsis and septic shock. The goal of this study is to measure the endotoxin activity of patients with severe sepsis and septic shock at certain time points, and furthermore, to compare the difference of endotoxin activity among different pathogens, infection source, and antibiotics. The study will enroll severe sepsis and septic shock patients. The endotoxin activity will be measured at certain time points according to the protocol.

DETAILED DESCRIPTION:
Endotoxin is the major mediator of gram-negative bacteria which cause the systemic inflammation and result in microcirculatory dysfunction, and it leads to multiple organ dysfunction and death in patients with severe sepsis and septic shock.

The goal of this study is to measure the endotoxin activity of patients with severe sepsis and septic shock at certain time points, and furthermore, to compare the difference of endotoxin activity among different pathogens, infection source, and antibiotics. The study will enroll severe sepsis and septic shock patients.

The endotoxin activity will be measured by Limulus Amebocyte Lysate (LAL) test. Limulus Amebocyte Lysate (LAL) test will be used to detect and quantify serum level of endotoxin. The critical component of the LAL reagents used in endotoxin tests is derived from blood cells (amebocytes) of the horseshoe crab, Limulus polyphemus. It contains the proteins of the blood clotting mechanism, which is triggered by endotoxins. LAL reagents are primarily used to test for endotoxins in injectable pharmaceuticals, biological products, and medical devices. They are also used in renal dialysis centers and a wide range of other applications. LAL tests are described in the Bacterial Endotoxins Test chapter in the United States Pharmacopeia (Chapter 85) and in the equivalent chapters in the European Pharmacopoeia (Chapter 2.6.14) and the Japanese Pharmacopoeia (Part I, General Tests, No. 6). We will adopt the chromogenic method as purchased from the Associates of Cape Cod Inc. (ACC). The LAL reagent is formulated with a synthetic substrate which gives a yellow color when acted upon by endotoxin activated enzyme. The test is read at 405 nm, usually in a microplate reader. The severity of multiple organ dysfunction and 28-day mortality will be followed up.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients with new onset of severe sepsis and septic shock
* Presence of at least 2 of the following conditions (These criteria should have occurred between 12 hours before or 6 hours after the onset of the qualifying first organ dysfunction)
* Fever or hypothermia (body temperature over 38 ℃ or under 36 ℃
* Tachycardia (heart rate > 90 bpm)
* Tachypnea (respiratory rate over 20 breaths/min or under mechanical ventilation)
* Leukocyte count more than 12,000 cells/mm3, less than 4,000 cells/mm3, or more than 10 % of immature form (band)

Exclusion Criteria:

Patient will be excluded if they

* are under 20 years old or older than 99 years old
* have suffered from severe sepsis or septic shock more than 24 hours
* are pregnant
* were treated with another medicine or device in the trial less than 30 days prior to the admission to this trial
* have received organ transplantation less than 1 years prior to this trial
* are terminally ill, for examples with metastasis, with a life expectancy of less than 30 days (certified by the attending physician)
* have already received other blood cleaning treatments, such as CVVH, HD, HF, and PE upon entry into the trial
* have chosen palliative care and signed Do Not Resuscitate sheet
* non-native speaker

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe sepsis and septic shock
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Endotoxin activity | baseline
  The endotoxin activity will be measured by Limulus Amebocyte Lysate (LAL) test. Limulus Amebocyte Lysate (LAL) test will be used to detect and quantify serum level of endotoxin.

SECONDARY OUTCOMES:
Change of endotoxin activity | At enrollment, 24h, 48h, and 72h
  Compare the change of endotoxin activity at different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, Ph.D., Principal Investigator — Department of Anesthesiology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan